CLINICAL TRIAL: NCT07398638
Title: A Phase Ib/II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Lisatoclax in Combination With R-CHOP or Pola-R-CHP in Patients With Previously Untreated DLBCL
Brief Title: Lisatoclax Plus R-CHOP or Pola-R-CHP in Untreated DLBCL: A Phase Ib/II Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-809
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Lisaftoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lisatoclax Combined with R-CHOP or Pola-R-CHP (Experimental): In Cohort 1, patients will receive standard-dose R-CHOP in combination with an initial dose of 400 mg of lisaftoclax. Each treatment cycle is 21 days. The lisaftoclax will be combined with R-CHOP at the RP2D dose level for an extension study.
  In Cohort 2, patients will receive standard-dose Pola-R-CHP in combination with an initial dose of 400 mg of lisaftoclax. Each treatment cycle is 21 days. The lisaftoclax will be combined with Pola-R-CHP at the RP2D dose level for an extension study.
  Interventions: Drug: R-CHOP; Drug: POLA-R-CHP; Drug: Lisaftoclax

INTERVENTIONS:
Drug: R-CHOP — Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
Drug: POLA-R-CHP — Polatuzumab vedotin, Rituximab, Cyclophosphamide, Doxorubicin, Prednisone
Drug: Lisaftoclax — Lisaftoclax (400 mg or 600 mg) is added from the second cycle of chemotherapy.

SUMMARY:
This is a prospective, multicenter, open-label Phase Ib/II clinical study designed to evaluate the safety, tolerability, preliminary efficacy, and pharmacokinetics of lisatoclax in combination with R-CHOP or Pola-R-CHP in patients with previously untreated diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in the clinical study; fully understand and be informed about the study and sign the Informed Consent Form (ICF); willing to comply with and capable of completing all trial procedures.
* 2. Diagnosed with DLBCL according to 2022 revised WHO lymphoma classification standards based on pathological diagnosis by the research center. For the dose-expansion phase, BCL-2 positivity (≥50% by IHC) is required.
* 3. Age 18-70 years.
* 4. No prior systemic anti-lymphoma therapy.
* 5. Adequate organ and bone marrow function.
* 6. At least one measurable or evaluable disease site according to the Lugano 2014 lymphoma efficacy evaluation criteria.
* 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

* 1. Lymphoma involvement in the central nervous system or meninges.
* 2. Active infections.
* 3. Uncontrolled clinical cardiac symptoms or diseases.
* 4. Currently using (or unable to stop at least one week prior to the first dose) a known CYP3A strong inducer or strong inhibitor.
* 5. Pregnant and lactating women, and subjects of childbearing age who do not want to use contraception.
* 6. History of Human Immunodeficiency Virus (HIV) infection and/or Acquired Immunodeficiency Syndrome (AIDS).
* 7. Patients with mental disorders or those unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) for Phase 1b | The first cycle (each cycle is 21 days) after lisaftoclax administration.
  To identify the DLT
Complete response rate (CRR) for Phase 2 | Up to 8 cycles (each cycle is 21 days)
  The proportion of patients who achieve complete response (CR)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 8 cycles (each cycle is 21 days)
  The proportion of patients who achieve complete response (CR) or partial response (PR)
Duration of Response (DOR) | Up to 5 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival (PFS) | Up to 5 years
  To investigate the preliminary anti-tumor efficacy
Overall survival (OS) | Up to 5 years
  To investigate the preliminary anti-tumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No